CLINICAL TRIAL: NCT03968965
Title: A Single-Center, Prospective Cohort Study of the Machine-vision Image Guided Surgery (MvIGS) Spine Navigation System
Brief Title: Evaluation of 3D Machine-vision Image Guided Surgery Spine Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 7D Surgical Inc. (Industry)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0328
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-03

CONDITIONS: Spinal Stenosis, Lumbar Region; Spondylolisthesis
Keywords: Image guided surgery; Computer-assisted surgery; Machine vision; Navigation; Image guidance; Spine; Lumbar spine
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: This is a single center, prospective, randomized cohort study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 3D MvIGS (Experimental): One, two and three-level posterior spine fusion surgery using bilateral pedicle screw instrumentation under 3D MvIGS intraoperative navigation guidance.
  Interventions: Device: 3D MvIGS Spine Navigation
- 2D Fluoroscopy (Other): One, two and three-level posterior spine fusion surgery using bilateral pedicle screw instrumentation under 2D fluoroscopy.
  Interventions: Other: 2D Fluoroscopy

INTERVENTIONS:
Device: 3D MvIGS Spine Navigation — The 7D Surgical MvIGS spine navigation system is for spatial positioning and orientation of surgical instruments during pedicle screw implantation in patients undergoing posterior fixation in single or multiple levels. The surgical light containing the machine vision cameras is the sole luminaire during image guided surgery.
  Arms: 3D MvIGS
Other: 2D Fluoroscopy — Pedicle screws will be placed using 2D fluoroscopy as the intraoperative imaging modality.
  Arms: 2D Fluoroscopy

SUMMARY:
This study assesses clinical outcomes following the use of the MvIGS spine navigation system for treatment of spinal stenosis and degenerative spondylolisthesis of the lumbar spine in adults. There will be separate study arms for cases utilizing the three-dimensional (3D) MvIGS spine navigation system and cases that utilize conventional two-dimensional (2D) fluoroscopy.

DETAILED DESCRIPTION:
This is a single center, randomized, prospective cohort study to comparatively evaluate the implementation of the MvIGS spine navigation system to conventional 2D fluoroscopy for pedicle screw fixation for the treatment of spinal stenosis with degenerative spondylolisthesis of the lumbar spine. Fluoroscopy and the MvIGS navigation system are both intraoperative imaging options available to aid spine surgeons.

Fluoroscopy uses X-rays to obtain images of patient anatomy. The MvIGS spine navigation system provides patient specific, high quality intraoperative imaging with no radiation exposure. After the spine is exposed, intraoperative images are obtained using visible light then registered to the patient's preoperative computed tomography scan. Use of the proprietary integrated surgical light with embedded tracking technology and Instant Flash™ registration allows for continuous and direct visualization of the surgical field without disturbing surgeon workflow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spinal stenosis of the lumbar spine with ≤ grade 2 degenerative spondylolisthesis
* Skeletally mature adults between the ages of 18-85 years at the time of surgery
* Has completed at least 6 months of conservative therapy
* Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Gross instability, defined as > 3 mm translational motion on flexion/extension studies
* Degenerative spondylolisthesis > grade 2
* Degenerative scoliosis > 10° at any level in lumbar spine
* Congenital lumbar spinal stenosis
* Endplate changes
* Visible change in disc height
* Radiographic confirmation of facet joint disease or degeneration
* Prior surgery at any lumbar level including the level being treated except for: Lamino/Foraminotomy, Microdiscectomy, IDET, and Percutaneous Discectomy
* Any evidence of a prior/current fracture, compromised vertebra, current or past trauma, or tumor at affected level or the spinous processes at the adjacent levels
* Requires destabilizing surgical decompression that adversely affects the functioning of the facets
* Cauda equina syndrome defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder dysfunction (bladder retention or incontinence)
* Significant peripheral neuropathy or acute denervation secondary to radiculopathy, caused by conditions other than spinal stenosis
* Significant peripheral vascular disease (diminished dorsalis pedis or tibial pulses)
* Morbid obesity, defined as BMI > 40 kg/m2
* Active systemic or local infection
* Active Hepatitis (receiving medical treatment within two years)
* Immunocompromised such as but not limited to Acquired Immunodeficiency Syndrome (AIDS), HIV infection, Severe Combined Immunodeficiency Syndrome, Thymic Hypoplasia
* Insulin dependent diabetes mellitus or any other medical condition(s) that would represent a significant increase in surgical risk or interfere with normal healing
* Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for > 1 month within last 12 months
* History of Paget's disease, osteomalacia, or any other metabolic bone disease
* Active malignancy. A patient with a history of any invasive malignancy (except nonmelanoma skin cancer), unless treated with curative intent and there has been no clinical signs or symptoms of the malignancy >5 years
* Involved in study of another investigational product that may affect outcome
* Women who are pregnant, lactating or anticipate becoming pregnant within 24 months post-surgery
* Patients who are incarcerated
* Worker's compensation cases
* Patients involved in active litigation relating to his/her spinal condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank P Cammisa, Jr., MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Guha D, Jakubovic R, Alotaibi NM, Klostranec JM, Saini S, Deorajh R, Gupta S, Fehlings MG, Mainprize TG, Yee A, Yang VXD. Optical Topographic Imaging for Spinal Intraoperative Three-Dimensional Navigation in Mini-Open Approaches: A Prospective Cohort Study of Initial Preclinical and Clinical Feasibility. World Neurosurg. 2019 May;125:e863-e872. doi: 10.1016/j.wneu.2019.01.201. Epub 2019 Feb 8. PMID 30743024
- [Background] Jakubovic R, Guha D, Gupta S, Lu M, Jivraj J, Standish BA, Leung MK, Mariampillai A, Lee K, Siegler P, Skowron P, Farooq H, Nguyen N, Alarcon J, Deorajh R, Ramjist J, Ford M, Howard P, Phan N, Costa LD, Heyn C, Tan G, George R, Cadotte DW, Mainprize T, Yee A, Yang VXD. High Speed, High Density Intraoperative 3D Optical Topographical Imaging with Efficient Registration to MRI and CT for Craniospinal Surgical Navigation. Sci Rep. 2018 Oct 5;8(1):14894. doi: 10.1038/s41598-018-32424-z. PMID 30291261

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Started | 32 | 32
Completed | 32 | 30
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants who did not complete the study, did not undergo a spinal procedure and were therefore, excluded from the baseline analysis population. The total number of baseline participants are those who underwent a spinal procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D MvIGS | 2D Fluoroscopy | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (12.5) | 63.9 (9.2) | 62.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 15 | 10 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Length of Operative Time
Description: Operative time determined by the official recorded operative notes
Time Frame: Data captured up to four hours after end of surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
minutes | 218 (37) | 218.5 (49)

2. Secondary Outcome: Length of Stay
Description: Length of hospital stay
Time Frame: Data captured upon patient discharge.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
Hours | 95.3 (34.7) | 98.4 (42.9)

3. Secondary Outcome: Estimated Blood Loss (EBL)
Description: Blood loss during surgery
Time Frame: During surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
mL | 408.6 (361.1) | 424.8 (211.8)

4. Secondary Outcome: Number of Misaligned Screws
Description: Number of screws that were misaligned as defined by discrepancies between the pilot hole and preoperative plan and final screw trajectory.
Time Frame: During hospital admission after surgery, an average of approximately 14 days
Measure: Number; unit: screws
Units Other Than Participants: Pedicle Screws
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
Number analyzed (Pedicle Screws) | 69 | 88
screws | 2 | 3

5. Secondary Outcome: Complications
Description: Number of reported complications (neurological deficits, dural tears, deep wound infections, etc.) while hospitalized
Time Frame: During hospital admission after surgery, an average of approximately 14 days
Measure: Number; unit: complications
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
complications | 0 | 0

6. Secondary Outcome: Measurement of Radiation Exposure
Description: Exposure measured by Dose Area Product (DAP)
Time Frame: During surgery
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
mGy | 10.3 (7.75) | 12.6 (7.30)

7. Secondary Outcome: Radiation Exposure Time
Description: Radiation exposure time
Time Frame: During surgery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 3D MvIGS | 2D Fluoroscopy
Number analyzed (Participants) | 32 | 30
seconds | 17.7 (11.23) | 18.7 (8.19)

ADVERSE EVENTS:
Time Frame: AEs were monitored throughout the study period, specifically, during surgery, immediately after surgery, and prior to patient discharge. Patients were monitored from discharge to their 6-month follow-up appointment, where any AEs during this timeframe will be assessed for a relationship to the patient's participation in the study, and if related, will be reported.
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study patient. All AEs will be recorded in this study. An AE can be any unfavorable and unintended sign, symptom, or disease regardless of the relationship to the product.
Arm/Group | 3D MvIGS | 2D Fluoroscopy
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03968965/Prot_SAP_000.pdf